CLINICAL TRIAL: NCT04104711
Title: The Outcomes of Home-Based Intervention to the Diabetics According to the Health Belief Model: A Randomized Controlled Trial
Brief Title: Home-Based Intervention to the Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilay AÇIL,PhD (Other)
Responsible Party: Sponsor-Investigator, Dilay AÇIL,PhD, Assistant Professor, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 970-GOA, 2014 / 07-20
Record Dates: First submitted 2019-09-16; First posted 2019-09-26 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2; Home Visit
Keywords: Diabetes; public health nursing; randomized controlled trials; chronic illness; Health Belief Model
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Chronic Disease | interventions — House Calls

STUDY DESIGN:
Intervention Model Description: During the first home visit, the participants in the intervention group were applied the data collection tools, and then nursing interventions in accordance with the subscales of the Health Belief Model by taking into account the individual differences of the participants. The nursing interventions were performed within the scope of the basic dimensions of diabetes management such as nutrition, exercise, medication management, etc. was also explained. Home visits were paid 3 times at 3-month intervals. After the home visits started, reminder messages supporting the home visit process were sent at two-week intervals. The participants in the control group were contacted 3 times at 3-month intervals through telephone calls, and were applied the data collection tools. At the end of the study, the participants in the control group were given health training and booklet was distributed to them.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home visits+Health education group (Experimental): Home visits were paid 3 times at 3-month intervals. After the home visits started, reminder messages supporting the home visit process were sent at two-week intervals.
  Nursing interventions were applied in accordance with the subscales of the Health Belief Model by taking into account the individual differences of the participants and were performed within the scope of the basic dimensions of diabetes management such as nutrition, exercise, medication management, oral care and foot care. In addition, the importance of annual monitoring of HBA1c, blood lipid, albumin/ creatinine levels, fundus examination, blood pressure monitoring, sleep hygiene, avoidance of smoking and alcohol was also explained.
  Interventions: Other: Home visits, health education
- No nursing intervention group (No Intervention): The participants in the control group who have standart care by other health services were contacted 3 times at 3-month intervals through telephone calls, and were applied the data collection tools only. They have no nursing intervention by the researcher.
  At the end of the study, for ethical statement the participants in the control group were given health training and the training booklet was distributed to them.

INTERVENTIONS:
Other: Home visits, health education
  Arms: Home visits+Health education group

SUMMARY:
Why is the research needed?

* This study reflects the complexity of the process that patients with diabetes are experiencing when staying at home away from the supervision of health professionals. In this context, there is a gap in the literature on home care of diabetes.
* The barriers, facilitators and the other perceptions that affect each diabetic's compliance with the disease-related recommendation are different. Nurses need to be aware of this.
* For this reason, according to the Health Belief Model, an original study was conducted to evaluate the nursing intervention program's results on patient care and cost-effectiveness in a home for supporting self-management of diabetic patients.

Hypotheses of the Study Patients with diabetes undergoing home-based nursing interventions in line with the Health Belief Model.

H1: have higher mean scores for the Health Belief Model Scale than the control group.

H2: have higher mean scores for the Self-Efficacy Scale than the control group. H3: have lower HbA1c levels than the control group. H4: have lower blood glucose levels (BGL) than the control group. H5: have lower blood pressure levels than the control group. H6: have lower BMI levels than the control group. H7: have fewer hospital admissions due to an acute or chronic complication than the control group.

H8: have a lower complication-related cost rate than the control group.

DETAILED DESCRIPTION:
Type of the study The study was conducted as an intervention (randomized controlled, single-blind) one.

Location and Time of the Study The study was carried out between January 2015 and March 2017 in three districts of İzmir, a province in the western part of Turkey.

The study population and sample While the patients with diabetes living in districts comprised the study population, the sample was selected from patients with type II diabetes registered to Family Health Centers.

According to the Consolidated Standards of Reporting Trials (CONSORT) recommended for randomized controlled studies, a randomization flow chart was established, and 2460 people with diabetes were assessed for compliance with diabetes. From the 1081 people with diabetes who met the inclusion criteria, the intervention, and control groups each to include 65 individuals were constructed using the "Research Randomizer" computer program. The study was completed with 81 people with diabetes (42 in the intervention group and 39 in the control group). Post hoc power analysis was performed using the G-Power Data Analysis program and the power of the study was determined as 100% at the 95% confidence interval and p = .05 significance level.

The participants were not told to which group they were assigned. Thus, the study was conducted as a single-blind study.

Training Booklet and Implementation Steps A booklet including information on nursing interventions for diabetes was prepared. The training booklet was based on the current literature and the results of the qualitative study conducted on the issue in the first step of the Ph.D. thesis. The booklet was revised in line with the opinions obtained from 5 professors who were experts in the field. The International Standard Book Number (978-975-441-462-2 ISBN) for the booklet was obtained by the Presidency of Dokuz Eylül University and published in the Dokuz Eylül University Press.

During the first home visit, the participants in the intervention group were applied the data collection tools, and then nursing interventions in accordance with the subscales of the Health Belief Model by taking into account the individual differences of the participants. The nursing interventions were performed within the scope of the basic dimensions of diabetes management such as nutrition, exercise, medication management, oral care, and foot care. In addition, the importance of annual monitoring of HBA1c, blood lipid, albumin/creatinine levels, fundus examination, blood pressure monitoring, sleep hygiene, avoidance of smoking and alcohol was also explained. Home visits were paid 3 times at 3-month intervals. After the home visits started, reminder messages supporting the home visit process were sent at two-week intervals.

The participants in the control group were contacted 3 times at 3-month intervals through telephone calls and were applied the data collection tools. At the end of the study, the participants in the control group were given health training at the Dokuz Eylül University Faculty of Nursing and the training booklet was distributed to them.

Analysis of the Data The study data were analyzed using numbers, percentages, the chi-square test, the test for the Signiﬁcance of the Difference Between Two Means, the Repeated Measures Multivariate Analysis of Variance, Bonferroni-adjusted t-test independent groups and multiple regression analysis in the Statistical Package for Social Sciences (SPSS) (23.0) program.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having Type 2 diabetes
* Not having diabetes-related complications
* Having a mobile phone to contact any time
* Living in the districts of Balçova, Narlıdere and Güzelbahçe

Exclusion Criteria:

* Having Type I diabetes
* Having been involved in a home care program previously
* Being illiterate in Turkish
* Having disabilities preventing the person from understanding others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Health Belief Model Scale in Patients with Diabetes | 6 month
  The Health Belief Model Scale was developed in China, the validity and reliability study of the Turkish version of the scale was conducted in 2007 and the Cronbach's alpha value was 0.72 and 0.90 respectively. The subscales of the scale were as follows: perceived Susceptibility (5 items), Perceived Severity (3 items), Perceived Benefits (7 items), Perceived Barriers (11 items) and Recommended health-related activities (10 items).
  The items of the scale are evaluated in a 5-point Likert scale, from 1 (I strongly disagree) to 5 (I strongly agree). Every subscale mean isdetermined by dividing the total points of all thesubscale items by the total number of items. The total scale score mean is calculated by dividing the totalpoints of all the items by the total number of items. A positive health belief of 4 points and above; a score below 4 is interpreted as a negative health belief.
Diabetes Management Self-Efficacy Scale for Patients with Type 2 Diabetes | 6 month
  Diabetes Management Self-Efficacy Scale was developed in 1999, the validity and reliability study of the Turkish version of the scale was conducted in 2001. The Cronbach's alpha value was 0.89 for both versions .The scale has 4 subscales: nutrition specific and weight, physical exercise, and blood sugar, nutrition general and medical treatment. The tool has 20 items. The items are in a 5-point Likert scale from 1 (absolutely no) to 5 (absolutely yes).The lowest possible score from the scale is 20, the highest is 100.
Fasting plasma glucose level (mg/dl) | 6 month
  The mean of plasma glucose level (milligram / deciliter) was used to compare patients' diabetic control and evaluate pre- and post-intervention values in the study process.
Postprandial glucose level (mg/dl) | 6 month
  The mean of postprandial glucose level (milligram / deciliter) was used to compare patients' diabetic control and evaluate pre- and post-intervention values in the study process.
Hemoglobin A1c level (%) | 6 month
  The mean of Hemoglobin A1c level (per cent) was used to compare patients' diabetic control by 3 months period and evaluate pre- and post-intervention values in the study process.
Body mass index (kg/m2) | 6 month
  Body mass index is important for metabolic control of diabetic patients. For this outcome weight and height of patients were measured. Then body mass index was calculated by the formula (weight (kilogram) / height (meter) x height (meter)). Body mass index were recorded kilogram/meter2.
Blood pressure level (mmHg) | 6 month
  Blood pressure levels were recorded milimeters mercury. Systolic and Diastolic Blood Pressure levels were measured both. This outcome is essential for macrovasculer complications.
Costs via frequency of complication-related hospital admissions | 6 month
  To calculate the cost of hospitalization for each patient, consumables (blood glucose measuring equipment, wound care products, wound cover, sterile gloves, catheter, urine bag, pen needle, infusion pump set) and time spent by the nurse (30 minutes for each patient) were determined. The cost of the time spent by the nurse was based on a new graduate nurse's salary and was calculated by using the formula '' salary ($)/ working time of May 2017 x 0.5 hours''.

OTHER OUTCOMES:
Sociodemographic and disease-related characteristics of patients with diabetes | First month
  This form includes questions about the sociodemographic and disease-related characteristics of patients with diabetes (age, sex, educational status, diagnose period, type of antidiabetic treatment, forgetfulness, glucose home monitoring, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Dilay AÇIL, Asst.Prof., Principal Investigator — Manisa Celal Bayar University; Zuhal BAHAR, Prof., Study Director — Koç University; Abdurrahman ÇÖMLEKÇİ, MD,Prof., Study Chair — Dokuz Eylul University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT04104711/Prot_SAP_000.pdf